CLINICAL TRIAL: NCT06891196
Title: Mixed-Methods Evaluation of Short-, Medium-, and Long-Term Outcomes Following Hip Treatment
Status: Active, not recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Emmanouil Grigoriou, Principal Investigator, Mayo Clinic
Other Study IDs: 24-012155
Record Dates: First submitted 2025-02-19; First posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Hip Dysplasia; Legg-Calvâe-Perthes Disease; Avascular Necrosis of Hip
MeSH Terms: conditions — Hip Dislocation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pediatric patients with hip conditions: Medical records and radiographs of patients who were treated for hip conditions at Mayo Clinic from 1975 to 2022 will be included in a retrospective chart review. Radiographic evaluations will include measurements of the neck-shaft angle, acetabular index, migration index, and other commonly used metrics.
  The prospective follow-up will include a subset of patients from the retrospective review, who will be complete long-term follow-up surveys.
  Interventions: Other: Long-term Follow-up Surveys

INTERVENTIONS:
Other: Long-term Follow-up Surveys — Patients will be given surveys, including validated PRO measures such as the Hip Disability and Osteoarthritis Outcomes Score (HOOS), Short-Form 12 (SF-12), Visual Analog Scale (VAS) for pain, and Marx activity scores.

SUMMARY:
This study, titled "Mixed-Methods Evaluation of Short-, Medium-, and Long-Term Outcomes Following Hip Treatment," aims to assess the long-term effectiveness of treatments for pediatric hip conditions, including hip dysplasia, Legg-Calve-Perthes disease, SCFE, and avascular necrosis.

DETAILED DESCRIPTION:
Conducted at Mayo Clinic, the study combines retrospective chart reviews and prospective follow-up to gather data on clinical outcomes, radiographic measures, and patient-reported outcomes (PROs) like functional status, pain, and quality of life.

The retrospective component analyzes records from 1975 to 2024, while the prospective component includes follow-up surveys using validated PRO measures (e.g., HOOS, SF-12, VAS). This study seeks to identify recurrence rates and complications associated with hip treatments, providing insights to improve future care standards for pediatric hip conditions. Data will be securely stored, with confidentiality maintained throughout.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18 seen for a concern of hip pathology at Mayo between 1975 and 2024
* Patients over 18 who can be contacted for follow-up and are willing to participate.

Exclusion Criteria:

* Patients presenting over age 18 for hip dysplasia
* Patients who are unwilling to complete follow up surveys.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients over the age of 18 seen for a concern of hip pathology at Mayo between 1975 and 2024.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
Revision surgery | 2 years
  Total number of patients who required revision surgery for pediatric hip conditions

SECONDARY OUTCOMES:
Change in neck-shaft angle measurement | Baseline, 2 years
  Radiographic measurement of the neck-shaft angle
Change in acetabular index | Baseline, 2 years
  Radiographic measurement of the acetabular index
Change in migration index | Baseline, 2 years
  Radiographic measurement of the migration index

CONTACTS AND LOCATIONS:
Overall Officials: Emmanouil Grigoriou, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No